CLINICAL TRIAL: NCT00794807
Title: A 12-Week Open-Label Followed by 4-Week Double-Blind Study to Determine the Safety and Efficacy of an Extended Course of Alefacept (LFA-3/IgG1 Fusion Protein) in Subjects With Chronic Plaque Psoriasis
Brief Title: Safety and Tolerability of Repeat Courses of IM Alefacept
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Biogen (Industry)
Responsible Party: Prof. W. Sterry, Dr. S. Philipp, Department of Dermatology and Allergy, Charite University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A Study of an Extended Regimen
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Last update posted 2008-11-20 (Estimated); Status verified 2008-11

CONDITIONS: Chronic Plaque Psoriasis
Keywords: Alefacept; Skin Diseases; Psoriasis; Skin Diseases, Papulosquamos; Therapeutic Uses; Dermatologic Agents
MeSH Terms: conditions — Skin Diseases; Psoriasis | interventions — Alefacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alefacept (Experimental)
  Interventions: Drug: Alefacept

INTERVENTIONS:
Drug: Alefacept — Alefacept=LFA-3/IgG1 fusion protein, once weekly, 15mg i.m.
  Other Names: LFA-3/IgG1 fusion protein

SUMMARY:
Previous Biogen studies have provided experience with the tolerability, immunogenicity, and efficacy of a single and multiple 12-week courses of therapy of alefacept. At this stage, experience in larger studies, as well as the FDA-approved labeling, is confined to treatment courses of 12 weeks. The purpose of the present study is to offer an extended course of therapy with alefacept.

DETAILED DESCRIPTION:
Twenty statistically matched patients (15 males, 5 females, aged between 28 and 70 years, median 50 years) with moderate to severe psoriasis (PASI: 7-36) were included in this study. They were treated with 15 mg alefacept i.m. weekly. Peripheral blood was taken prior to first alefacept application and then weekly until week five and thereafter every second week, until the end of treatment at week 13. At the same time points severity of disease and thereby possible reduction of symptoms was evaluated applying the PASI. Investigators analysing the samples were blinded to the outcome of the study. The protocol concerning human subjects was approved by the ethics commission of the Charité University Medicine Berlin Campus Mitte, Germany .

ELIGIBILITY:
Inclusion Criteria:

1. Must give written informed consent.
2. Must require systemic therapy or phototherapy for their psoriasis, as determined by the investigator prior to Visit 1.

Exclusion Criteria:

1. Female subjects who are not postmenopausal for at least 1 year, surgically sterile, or willing to practice effective contraception during the study. Nursing mothers, pregnant women and women planning to become pregnant while on study are to be excluded.
2. Current enrollment in any investigational study in which the subject is receiving any type of drug, biologic, or non-drug therapy (participation in registry-type studies is allowed).
3. Serious local infection (e.g., abscess) or systemic infection (e.g., pneumonia, septicemia) within the 3 months prior to the first dose of investigational drug.
4. Any subject whose CD4+ lymphocyte count at study entry is less than 404 cells/mm3.
5. Treatment with another investigational drug or approved therapy for investigational use within 28 days prior to investigational drug administration.
6. Treatment with systemic retinoids, systemic steroids, methotrexate, cyclosporine, azathioprine, thioguanine or other systemic immunosuppressant agents within the 28 days prior to investigational drug administration.
7. Phototherapy, including Ultraviolet B (UVB) and Psoralen + Ultraviolet A (PUVA), within 28 days prior to investigational drug administration.
8. Known HIV+, known viral Hepatitis infection, known tuberculosis infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-02; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Safety of an extended courses of alefacept when administered to subjects with chronic plaque psoriasis. Safety parameters: Physical examinations; vital signs; infections; blood test: lymphocyte subset analysis (CD4+); and adverse events. | 12 + 4 weeks

SECONDARY OUTCOMES:
Efficacy of an extended course of alefacept when administered to subjects with chronic plaque psoriasis: Time to requirement of additional systemic therapies, Psoriasis Area and Severity Index (PASI); Physician Global Assessment (PGA). | 12 + 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wolfram Sterry, Prof. M.D., Study Director — Department of Dermatology and Allergy, Charité-Universitaetsmedizin Berlin
Locations (1):
- Psoriasis Study center, The interdisciplinary group of Molecular Immunopathology, Berlin, State of Berlin, Germany